CLINICAL TRIAL: NCT05253781
Title: Low Dose Aspirin for Preventing Intrauterine Growth Restriction and Preeclampsia in Sickle Cell Pregnancy (PIPSICKLE): a Randomized Controlled Trial
Brief Title: Low Dose Aspirin for Preventing Intrauterine Growth Restriction and Preeclampsia in Sickle Cell Pregnancy (PIPSICKLE)
Acronym: PIPSICKLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Lagos, Nigeria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PACTR202001787519553; 2021-002867-23 (EudraCT Number)
Record Dates: First submitted 2021-12-14; First posted 2022-02-24 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Intrauterine Growth Restriction; Preeclampsia; Sickle Cell Disease; Pregnancy Complications
Keywords: Sickle cell disease; Low dose aspirin; Preeclampsia; Intrauterine growth restriction (IUGR); Pregnancy complications
MeSH Terms: conditions — Fetal Growth Retardation; Pre-Eclampsia; Anemia, Sickle Cell; Pregnancy Complications | interventions — Aspirin; Basigin

STUDY DESIGN:
Intervention Model Description: The clinical trial aspect is a multi-centre parallel, double blind, superiority randomized controlled trial, with women allocated in a 1:1 ratio. Participants are randomized into two groups. One group receiving low dose aspirin (LAD) 100mg daily from 12 weeks or from enrollment to 36 weeks gestational age. The second group receives a placebo tablet that looks exactly like the LAD in colour, size and shape also one tablet daily from 12 weeks or from enrollment to 36 weeks gestational age.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind design. An unblinded pharmacist does the drug packaging and has the code for drug identification. All other members of the research team and patients are blinded and do not know what each drug is.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Low dose aspirin (LDA) group will receive 100mg aspirin daily taken at once just before bedtime from 12 weeks gestational age or enrollment till 36 weeks gestational age.
  Interventions: Drug: Low-dose aspirin
- Control (Placebo Comparator): Placebo group will receive one tablet of the placebo which has same shape, size, thickness and colour as the LDA daily taken at once just before bedtime from 12 weeks gestational age or enrollment till 36 weeks gestational age.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Low-dose aspirin — Low dose aspirin (LDA) group will receive 100mg aspirin daily taken at once just before bedtime from 12 weeks gestational age or enrollment till 36 weeks gestational age.
  Other Names: Emprin
  Arms: Intervention
Other: Placebo — Placebo group will receive one tablet of the placebo which has same shape, size, thickness and colour as the LDA daily taken at once just before bedtime from 12 weeks gestational age or enrollment till 36 weeks gestational age.
  Other Names: Emprin placebo
  Arms: Control

SUMMARY:
Pregnancy in sickle cell disease (SCD) is fraught with many complications including preeclampsia (PE) and intrauterine growth restriction (IUGR). Previously, the investigators found an abnormality in prostacyclin-thromboxane ratio in sickle cell pregnant women, a situation that is also found in non-sickle pregnancies with PE and unexplained IUGR. Low dose aspirin (LDA) has been found to reduce the incidence of PE and IUGR in high-risk women due to its reduction of vasoconstrictor thromboxane whilst sparing prostacyclin, in effect "correcting" the ratio. It has been found to be safe for use in pregnancy and is recommended in obstetric guidelines for this use but has not been tested in sickle cell pregnancy. The investigators hypothesize that LDA would reduce the incidence of IUGR and PE in pregnant haemoglobin (Hb)SS women. The investigators also plan to build a machine-learning model to predict severe maternal outcomes in them.

The investigators propose a multi-site, randomized, controlled, double blind trial comparing a daily dose of 100mg aspirin with placebo, from 12 - 28 weeks gestation until 36 weeks. The study sites are three teaching hospitals in Lagos and Ile-Ife, and twelve general hospitals and one federal medical centre within Lagos state, with the coordinating centre at the College of Medicine, University of Lagos (CMUL), Idi-Araba, Lagos. A total of 476 eligible pregnant HbSS and HbSC women will be recruited consecutively and randomly assigned to either group using a web-based app, sealed envelope. Each study group will comprise 238 pregnant women with SCD.

All participants will be followed from recruitment till six weeks postpartum. They will have their body weight, blood pressure and haematocrit checked at each antenatal visit. Their full blood count, vital signs and oxygen saturation will be checked and recorded at each visit. Primary outcome measure will be birth weight below 10th centile for gestational age on INTERGROWTH 21 birthweight charts, and incidence of miscarriage or perinatal death. Analysis will be by intention to treat, and the main treatment effects will be quantified by relative risk with 95% confidence intervals, at a 5% significance level. The investigators plan to develop a prediction model to predict the risk of complications in these women using machine learning. The prediction outcome will be severe maternal outcomes comprising maternal near miss or death.

DETAILED DESCRIPTION:
STUDY RATIONALE Sickle cell disease (SCD) especially in pregnancy poses great burden and is thus designated a global public health problem by World Health Organization (WHO) and United Nations. In Nigeria, many SCD women die because of pregnancy complications. The physiological changes in pregnancy aggravate the severity of pregnancy complications in women with SCD. Maternal mortality ratio and perinatal mortality rate in Nigeria till date has remained high. Hypertensive disorders of pregnancy, which includes preeclampsia (PE) is a leading cause of maternal death and intrauterine growth restriction (IUGR) and low birth weight (LBW) are leading causes of perinatal deaths. Pregnancy outcomes in women with SCD follows a variable course and it is thus difficult to identify those who will develop complications during pregnancy. There is thus a need to develop cost-effective strategies to prevent complications in this category of women. However very few randomized controlled trials address their management, and guidelines for their treatment are supported by low quality evidence. Low dose aspirin (LDA) has been found to be beneficial in prevention of preeclampsia in non-SCD pregnant women. The NICE guideline lists several risk factors for preeclampsia for which LDA is recommended but no mention is made of women with SCD who are known to be at high risk of preeclampsia. This research is therefore targeted at determining if drugs such as LDA may be beneficial in reducing the contributions of this genetic condition to maternal and perinatal deaths in a low resource setting like ours, consequently saving economic as well as physical resources.

The aim of this clinical trial is to determine whether daily administration of 100mg LDA from 12 - 28 weeks of gestation till 36 weeks, reduces the risk of IUGR, PE, perinatal deaths or miscarriages and other complications (sickling and non-sickling related) in pregnant HbSS women compared with the use of placebo.

OBJECTIVES

1. To determine the effect of the use of LDA during pregnancy in HbSS and HbSC women on the risk of IUGR, perinatal death or miscarriage.
2. To determine the effect of the use of LDA during pregnancy in HbSS and HbSC women on the risk of other maternal complications including PE, preterm delivery, number of vaso-occlusive crises, need for blood transfusion, urinary tract infections, respiratory tract infections, acute chest syndrome, retained placenta, placental abruption, and vaginal bleeding.

METHODOLOGY Study design A multi-centre parallel, double blind, superiority randomized controlled trial, with women allocated in a 1:1 ratio into two groups, namely low dose aspirin (LDA) group and placebo group.

Settings and locations Study sites include 3 Teaching Hospitals in Lagos and Ife, Osun State, 12 General Hospitals in Lagos and 1 Federal Medical Centre within Lagos State. The coordinating centre is College of Medicine, University of Lagos (CMUL), Lagos, Nigeria.

Sample size Using the formula for proportions in superiority parallel trials and assuming an incidence of IUGR of 20% in SCD and expecting a 50% IUGR reduction with the use of LDA as detected by Bujold et al, 476 women in total (238 women per group) was calculated to give this study a 90% power of detecting a decrease in IUGR at the 5% significance level and allowing for 20% attrition.

Enrolment and data collection Each woman at 12 to 28 weeks gestation who self-reports or is found to have SCD on routine haemoglobin genotype testing, will have a confirmatory haemoglobin electrophoresis done. This is to have a uniform diagnosis and to be certain of the exact sickle cell phenotype. Every woman with haemoglobin SS or SC that fits the eligibility criteria and gives informed consent will be consecutively recruited. They will be randomized into either LDA group or placebo group using a web-based software, Sealed envelope, in a 1:1 ratio in blocks stratified according to centre. Only an unblinded pharmacist, will be aware of the actual codes and she will not be in contact with any of the study participants. Those in the LDA group will receive 100mg aspirin daily taken at once just before bedtime while those in the placebo group will receive a tablet that looks like the active drug in terms of size and thickness. The drugs will be continued till 36 weeks or delivery, whichever comes earlier. The women will have their haemoglobin fraction assayed by HPLC, mid-stream urine for microscopy, culture and sensitivity done and full blood count will be done at enrolment.

The women will be seen 2 - 4 weekly in the antenatal clinic up till 28 weeks and then weekly thereafter till delivery. Their body weight, blood pressures, haemoglobin concentration and urinalysis for protein and glucose will be measured at every visit. If proteinuria of ≥1+ (≥30mg/dl) is recorded in a participant with elevated blood pressure (hypertension), urine specimen will be collected for urinary protein to creatinine ratio estimation (UPCR) to confirm if proteinuria is significant, a value of 30mg/mmol will be considered significant. Their full blood count will be repeated at delivery. They will have an ultrasound scan at 20 weeks. Their oxygen saturation will be monitored in addition to other vital signs such as pulse rate, blood pressure, temperature, and respiratory rates whenever they are admitted to the hospital. At delivery, the babies will be weighed naked to detect low birth weight based on WHO INTERGROWTH-21st Chart. Placenta biopsies will be taken for histology to identify abnormalities that might be associated with some pregnancy complications such as PE and IUGR.

Adverse events will be recorded on the adverse event CRF as any symptom that starts or worsens after study drugs have been commenced. The severity (mild, moderate, severe) of adverse drug event, relationship to the study drug (suspected/not suspected), duration (start and end dates or if continuing at final exam) and whether it constitutes a serious adverse event (SAE) will be recorded at each visit. Pill count will be done at each visit. Reminder messages and call will be made to remind participants to take their drugs and to make their appointments. Participants who miss a visit will be tracked to their houses, if necessary, as a strategy to minimize loss to follow up. The participants were followed up till six weeks postpartum.

Data analysis plan Data analysis will be by intention-to-treat. Categorical variables will be expressed as frequencies and percentages. For continuous variables, a Shapiro-Wilk test of normality will be performed, and normally distributed data will be presented as means ± SD, while non-normally distributed data will be presented as median and interquartile range (IQR). Risk of occurrence of IUGR, perinatal death and other key outcome variables will be computed and compared in both groups. A multivariate regression analysis will be performed to determine the odds of each of the key outcomes among women who received the intervention with respect to those who did not, after controlling for common confounders. This will be presented as regression coefficients and their 95% confidence intervals. Level of significance will be set at 5%. Post-regression analysis will be performed to determine the goodness-of-fit of the final model. STATA version15.0 (Stata Corp LP, College Station, TX, USA) will be used for statistical analysis.

QUALITY CONTROL AND DATA MANAGEMENT Data will be double entered with assigned codes. Data will be captured in electronic case report forms (CRF) at various patient visit types and uploaded real time to the central server after being checked by site coordinators. They will follow guidelines specified in the SOP developed by the Data handling and communications committee for data collection, data entry, and transmission, data compilation and management and data quality and security.

ETHICAL AND ENVIRONMENTAL CONSIDERATIONS The clinical trial is registered in Pan African Clinical Trials Registry (PACTR202001787519553) and has ethical approvals from Health Research and Ethics committees of Lagos University Teaching Hospital, Idi-Araba (ADM/DST/HREC/APP/3301), Lagos State University Teaching Hospital, LASUTH (LREC/06/10/1318), Federal Medical Centre, Ebute Metta (FMCEB/RET/0052), Health Service Commission of Lagos State (LSHSC/2222/VOLIII), and National Health Research and Ethics Committee (NHREC/01/01/2007-04/12/2020).

Personal data of participants will be kept strictly confidential. All data will be stored securely in a central electronic database by the PI who will be the only one who will have access to the data of all participants collated centrally. The statistician will be granted access to the electronic database during statistical analysis or at any other time the PI might require her to review the data. None of the women will be made to pay for any aspect of the study as trial drugs and investigations will be offered at no cost. All participants will receive their routine medications (malaria prophylaxis, tetanus toxoid prophylaxis and folic acid supplementation) normally. Free malaria prophylaxis and folic acid will be given to them all through pregnancy as an incentive for participating in the research. Participants will have autonomy to participate and a right to withdraw from the study if they wish to do so. All participants will enjoy equal rights and quality care all through the duration of the research. Environmental issues are not applicable to this study.

MONITORING AND EVALUATION MECHANISM The M &E mechanism will include an Administrative Core consisting of the PI and a full-time project coordinator who will provide administrative oversight and management of the research study and coordinate all internal and external meetings of investigators and staff. A Steering Committee comprising PI, all co-investigators, site coordinators and a patient representative will be constituted, and will monitor project progress and ensure compliance with regulatory, fiscal, and reporting requirements. Clinical Trial Monitors who will be responsible for trial monitoring will also be appointed. A Data and Safety Monitoring Board (DSMB) will also be constituted.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Singleton fetus
* Women whose genotypes are Haemoglobin SS or SC.
* 28 weeks gestation or less at recruitment, estimated from the last menstrual period or by an early ultrasound scan.

Exclusion Criteria:

* Women with associated medical conditions in pregnancy e.g., HIV infection, diabetes mellitus, hypertension, renal disease, sickle nephropathy
* Multiple pregnancy
* Hypersensitivity to aspirin
* History of blood transfusion in the last 3 months
* Women who participated in the PIPSICKLE trial during their previous pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on self-representation of gender identity and confirmed pregnancy.
Enrollment: 476 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Number of babies with birth weight below 10th centile for gestational age on the WHO INTERGROWTH-21st birthweight charts, stillbirth or fetal death or miscarriages divided by the total number of babies delivered. | up to seven days after delivery.
  Intrauterine growth restriction, perinatal death or miscarriage as a composite outcome.

SECONDARY OUTCOMES:
Number of participants who will develop preeclampsia defined as hypertension and significant proteinuria after 20 weeks gestational age divided by the total number of participants. | To be measured from date of randomization if greater than 20 weeks up till 6 weeks post-delivery if present
  Number of participants who will develop preeclampsia defined as hypertension and significant proteinuria (1+ proteinuria (≥30 mg dl-1) on two occasions at least 4 hours apart without any evidence of a urinary tract infection or protein 2+ or more on dipstick or urinary protein creatinine ratio >300mg/g) after 20 weeks gestational age divided by the total number of participants.
Number of women that die at any gestational age during pregnancy or within 42 days after delivery from any cause arising from the pregnancy or its management but not from incidental or accidental causes, divided by the total number of participants. | To be measured from randomization until date of death or 6 weeks post-delivery whichever comes first,
  maternal death
Number of women delivered before 37 weeks gestational age divided by the total number of participants randomized. | up to preterm delivery.
  preterm delivery
Number of participants who will develop thromboembolism divided by the total number of participants. | To be measured from randomization until date of death or 6 weeks post-delivery whichever comes first,
  Thromboembolism
Number of babies who died from 28 weeks gestational age up to seven days post delivery (comprising all still births and early neonatal deaths divided by total births reported as percentage. | from 28 weeks gestational age till seven days post delivery
  Perinatal death.
Mean number of sickle cell crises in participants in each arm. | from enrolment till six weeks postpartum.
  Number of sickle cell crisis.
Number requiring blood transfusion. | from enrolment till six weeks postpartum.
  Need for blood transfusion per arm.
Number of women with urinary tract infection in each arm. | from enrolment till six weeks postpartum.
  Urinary tract infection.
Number of women with lower respiratory tract infection (pneumonia) in each arm. | from enrolment till six weeks postpartum.
  Lower respiratory tract infection (pneumonia).
Number of women with acute chest syndrome in each arm. | from enrolment till six weeks postpartum.
  Acute chest syndrome.
Number of women with retained placenta in each arm. | from enrolment till six weeks postpartum.
  Retained placenta.
Number of women with placenta abruptio in each arm. | from enrolment till six weeks postpartum.
  Abruptio placenta
Number of participants with adverse drug events. | from enrolment 36 weeks gestational age.
  Adverse drugs events like vaginal bleeding, epigastric pain and heartburn.

CONTACTS AND LOCATIONS:
Overall Officials: Bosede B Afolabi, DM (Nott), Principal Investigator — College of Medicine, University of Lagos
Locations (16):
- Nigeria (16):
  - Ajeromi General Hospital, Ajegunle, Lagos State, Ajegunle, Lagos
  - Federal Medical Centre, Ebute Metta, Lagos State, Ebute-Metta, Lagos
  - Lagos University Teaching Hospital, Idi Araba, Lagos
  - Alimosho General Hospital, Igando, Lagos State, Igando, Lagos
  - Lagos State University Teaching Hospital (LASUTH, Ikeja, Lagos
  - General Hospital, Ikorodu, Lagos State, Ikorodu, Lagos
  - General Hospital, Isolo, Lagos State, Isolo, Lagos
  - General Hospital, Somolu, Lagos State, Somolu, Lagos
  - Randle General Hospital, Surulere, Lagos State, Surulere, Lagos
  - Obafemi Awolowo University Teaching Hospital OAUTH), Ife, Osun State, Ile-Ife, Osun State
  - Lagos Island Maternity Hospital, Lagos, Lagos
  - General Hospital, Gbagada, Lagos State, Lagos
  - General Hospital, Ibeju-Lekki, Lagos State, Lagos
  - General Hospital, Ifako Ijaiye, Lagos State, Lagos
  - General Hospital, Orile-Agege, Lagos State, Lagos
  - Mother and Child Centre, Amuwo-Odofin, Lagos, Lagos

IPD SHARING:
Plan to Share IPD: Yes
We will store the data and deposit it in 'Open Science Framework', after approval is obtained from the ethics committee. We will also provide metadata along with the data to describe it. No patient identifier will be included in data shared. Potential new users may access our data including the metadata on the 'Open Science Framework'. We will share the data at the time of publication of our first paper. The assigned DOI number, the OSF website details and our approach to data sharing will be included as an appendix to all publications emanating from this research to facilitate accessibility to our data and metadata. We will also share these at any conference presentation both international and local, and also on our study website to facilitate access to it by other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD and supporting information will be made available at the time of first paper publication and will be made available for a period of 2 years
Access Criteria: 1. Governance of access The principal investigator will bear overall responsibility for this data and will be responsible for deciding whether to supply research data to a potential new user. The CMUL HREC will provide an independent oversight function. 2. The study team's exclusive use of the data Data will be made available at the time of publication, at the latest. Depending on the nature of the data itself, data may be made available earlier, either on an individual basis to interested researchers and/or potential new collaborators. 3. Restrictions or delays to sharing, with planned actions to limit such restrictions We will ensure that our informed consent forms clearly spell out and seek consent for future data sharing. 4. Regulation of responsibilities of users All external users will sign and be bound by our data sharing agreements and will not be allowed to use the data for reasons other than stated in their application.

REFERENCES:
- [Background] WHO. Sickle-cell Anaemia Report by the Secretariat. World Health Organisation. Fifty-ninth World Health Assembly; 2006a. Report No.: A59/9 Contract No.: Provisional agenda item 11.4.
- [Background] Chakravorty S, Williams TN. Sickle cell disease: a neglected chronic disease of increasing global health importance. Arch Dis Child. 2015 Jan;100(1):48-53. doi: 10.1136/archdischild-2013-303773. Epub 2014 Sep 19. PMID 25239949
- [Background] Yawn BP, Buchanan GR, Afenyi-Annan AN, Ballas SK, Hassell KL, James AH, Jordan L, Lanzkron SM, Lottenberg R, Savage WJ, Tanabe PJ, Ware RE, Murad MH, Goldsmith JC, Ortiz E, Fulwood R, Horton A, John-Sowah J. Management of sickle cell disease: summary of the 2014 evidence-based report by expert panel members. JAMA. 2014 Sep 10;312(10):1033-48. doi: 10.1001/jama.2014.10517. PMID 25203083
- [Background] Rees DC, Williams TN, Gladwin MT. Sickle-cell disease. Lancet. 2010 Dec 11;376(9757):2018-31. doi: 10.1016/S0140-6736(10)61029-X. Epub 2010 Dec 3. PMID 21131035
- [Background] Oteng-Ntim E, Ayensah B, Knight M, Howard J. Pregnancy outcome in patients with sickle cell disease in the UK--a national cohort study comparing sickle cell anaemia (HbSS) with HbSC disease. Br J Haematol. 2015 Apr;169(1):129-37. doi: 10.1111/bjh.13270. Epub 2014 Dec 18. PMID 25522142
- [Background] Villers MS, Jamison MG, De Castro LM, James AH. Morbidity associated with sickle cell disease in pregnancy. Am J Obstet Gynecol. 2008 Aug;199(2):125.e1-5. doi: 10.1016/j.ajog.2008.04.016. Epub 2008 Jun 4. PMID 18533123
- [Background] Afolabi BB, Iwuala NC, Iwuala IC, Ogedengbe OK. Morbidity and mortality in sickle cell pregnancies in Lagos, Nigeria: a case control study. J Obstet Gynaecol. 2009 Feb;29(2):104-6. doi: 10.1080/01443610802667112. PMID 19274540
- [Background] Say L, Souza JP, Pattinson RC; WHO working group on Maternal Mortality and Morbidity classifications. Maternal near miss--towards a standard tool for monitoring quality of maternal health care. Best Pract Res Clin Obstet Gynaecol. 2009 Jun;23(3):287-96. doi: 10.1016/j.bpobgyn.2009.01.007. Epub 2009 Mar 19. PMID 19303368
- [Background] Ellis RJ, Wang Z, Genes N, Ma'ayan A. Predicting opioid dependence from electronic health records with machine learning. BioData Min. 2019 Jan 29;12:3. doi: 10.1186/s13040-019-0193-0. eCollection 2019. PMID 30728857
- [Background] Yang F, Banerjee T, Narine K, Shah N. Improving Pain Management in Patients with Sickle Cell Disease from Physiological Measures Using Machine Learning Techniques. Smart Health (Amst). 2018 Jun;7-8:48-59. doi: 10.1016/j.smhl.2018.01.002. Epub 2018 Feb 2. PMID 30906841
- [Background] Obilade OA, Akanmu AS, Broughton Pipkin F, Afolabi BB. Prostacyclin, thromboxane and glomerular filtration rate are abnormal in sickle cell pregnancy. PLoS One. 2017 Sep 7;12(9):e0184345. doi: 10.1371/journal.pone.0184345. eCollection 2017. PMID 28880908
- [Background] Lewis DF, Canzoneri BJ, Gu Y, Zhao S, Wang Y. Maternal levels of prostacyclin, thromboxane, ICAM, and VCAM in normal and preeclamptic pregnancies. Am J Reprod Immunol. 2010 Dec;64(6):376-83. doi: 10.1111/j.1600-0897.2010.00861.x. PMID 20482519
- [Background] Duley L, Henderson-Smart DJ, Knight M, King JF. Antiplatelet agents for preventing pre-eclampsia and its complications. Cochrane Database Syst Rev. 2004;(1):CD004659. doi: 10.1002/14651858.CD004659. PMID 14974075
- [Background] Moore GS, Allshouse AA, Post AL, Galan HL, Heyborne KD. Early initiation of low-dose aspirin for reduction in preeclampsia risk in high-risk women: a secondary analysis of the MFMU High-Risk Aspirin Study. J Perinatol. 2015 May;35(5):328-31. doi: 10.1038/jp.2014.214. Epub 2014 Dec 4. PMID 25474553
- [Background] RCOG. Management of Sickle Cell Disease in Pregnancy. Royal College of Obstetricians and Gynaecologists Green-top Guideline. 2011:1-20.
- [Background] Boafor TK, Olayemi E, Galadanci N, Hayfron-Benjamin C, Dei-Adomakoh Y, Segbefia C, Kassim AA, Aliyu MH, Galadanci H, Tuuli MG, Rodeghier M, DeBaun MR, Oppong SA. Pregnancy outcomes in women with sickle-cell disease in low and high income countries: a systematic review and meta-analysis. BJOG. 2016 Apr;123(5):691-8. doi: 10.1111/1471-0528.13786. Epub 2015 Dec 15. PMID 26667608
- [Background] Afolabi B. Plasma volume in normal and sickle cell pregnancy. United Kingdom: University of Nottingham; 2011.
- [Background] Afolabi BB, Oladipo OO, Akanmu AS, Abudu OO, Sofola OA, Broughton Pipkin F. Volume regulatory hormones and plasma volume in pregnant women with sickle cell disorder. J Renin Angiotensin Aldosterone Syst. 2016 Sep 27;17(3):1470320316670444. doi: 10.1177/1470320316670444. Print 2016 Jul. PMID 27678389
- [Background] Tohgi H, Konno S, Tamura K, Kimura B, Kawano K. Effects of low-to-high doses of aspirin on platelet aggregability and metabolites of thromboxane A2 and prostacyclin. Stroke. 1992 Oct;23(10):1400-3. doi: 10.1161/01.str.23.10.1400. PMID 1412574
- [Background] Capone ML, Tacconelli S, Sciulli MG, Grana M, Ricciotti E, Minuz P, Di Gregorio P, Merciaro G, Patrono C, Patrignani P. Clinical pharmacology of platelet, monocyte, and vascular cyclooxygenase inhibition by naproxen and low-dose aspirin in healthy subjects. Circulation. 2004 Mar 30;109(12):1468-71. doi: 10.1161/01.CIR.0000124715.27937.78. Epub 2004 Mar 22. PMID 15037526
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] Henderson JT, Whitlock EP, O'Connor E, Senger CA, Thompson JH, Rowland MG. Low-dose aspirin for prevention of morbidity and mortality from preeclampsia: a systematic evidence review for the U.S. Preventive Services Task Force. Ann Intern Med. 2014 May 20;160(10):695-703. doi: 10.7326/M13-2844. PMID 24711050
- [Background] NICE. Hypertension in pregnancy: the management of hypertensive disorders during pregnancy. National Institute for Health and Clinical Excellence Clinical Guideline. 2010;107:1-47.
- [Background] Ahrens KA, Silver RM, Mumford SL, Sjaarda LA, Perkins NJ, Wactawski-Wende J, Galai N, Townsend JM, Lynch AM, Lesher LL, Faraggi D, Zarek S, Schisterman EF. Complications and Safety of Preconception Low-Dose Aspirin Among Women With Prior Pregnancy Losses. Obstet Gynecol. 2016 Apr;127(4):689-698. doi: 10.1097/AOG.0000000000001301. PMID 26959198
- [Background] Xu TT, Zhou F, Deng CY, Huang GQ, Li JK, Wang XD. Low-Dose Aspirin for Preventing Preeclampsia and Its Complications: A Meta-Analysis. J Clin Hypertens (Greenwich). 2015 Jul;17(7):567-73. doi: 10.1111/jch.12541. Epub 2015 Apr 2. PMID 25833349
- [Background] Mone F, Mulcahy C, McParland P, McAuliffe FM. Should we recommend universal aspirin for all pregnant women? Am J Obstet Gynecol. 2017 Feb;216(2):141.e1-141.e5. doi: 10.1016/j.ajog.2016.09.086. Epub 2016 Sep 20. PMID 27659212
- [Background] Resende Cardoso PS, Lopes Pessoa de Aguiar RA, Viana MB. Clinical complications in pregnant women with sickle cell disease: prospective study of factors predicting maternal death or near miss. Rev Bras Hematol Hemoter. 2014 Jul-Aug;36(4):256-63. doi: 10.1016/j.bjhh.2014.05.007. Epub 2014 May 29. PMID 25031164
- [Background] Al-Farsi SH, Al-Riyami NM, Al-Khabori MK, Al-Hunaini MN. Maternal complications and the association with baseline variables in pregnant women with sickle cell disease. Hemoglobin. 2013;37(3):219-26. doi: 10.3109/03630269.2013.780249. Epub 2013 Apr 17. PMID 23590330
- [Background] Jhee JH, Lee S, Park Y, Lee SE, Kim YA, Kang SW, Kwon JY, Park JT. Prediction model development of late-onset preeclampsia using machine learning-based methods. PLoS One. 2019 Aug 23;14(8):e0221202. doi: 10.1371/journal.pone.0221202. eCollection 2019. PMID 31442238
- [Background] Brown MA, Lindheimer MD, de Swiet M, Van Assche A, Moutquin JM. The classification and diagnosis of the hypertensive disorders of pregnancy: statement from the International Society for the Study of Hypertension in Pregnancy (ISSHP). Hypertens Pregnancy. 2001;20(1):IX-XIV. doi: 10.1081/PRG-100104165. No abstract available. PMID 12044323
- [Background] Nwabuko OC, Okoh DA, Iyalla C, Omunakwe H. Prevalence of sickle cell disease among pregnant women in a tertiary health center in south-south Nigeria. Sub-Saharan Afr J Med. 2016; 3:132-6.
- [Background] Olugbenga AO. Managing sickle cell disease in pregnancy, the success, and the challenges: Our experience in a semi-urban tertiary health-care facility, Southwest, Nigeria. Trop J Obstet Gynaecol 2018; 35:342-7.
- [Background] Babah OA, Aderolu MB, Oluwole AA, Afolabi BB. Towards zero mortality in sickle cell pregnancy: A prospective study comparing haemoglobin SS and AA women in Lagos, Nigeria. Niger Postgrad Med J. 2019 Jan-Mar;26(1):1-7. doi: 10.4103/npmj.npmj_177_18. PMID 30860192
- [Background] United Nations, Department of Economic and Social Affairs, Population Division (2018). World Urbanization Prospects: The 2018 Revision, Online Edition. https://population.un.org/wup/Download/
- [Background] Al Jama FE, Gasem T, Burshaid S, Rahman J, Al Suleiman SA, Rahman MS. Pregnancy outcome in patients with homozygous sickle cell disease in a university hospital, Eastern Saudi Arabia. Arch Gynecol Obstet. 2009 Nov;280(5):793-7. doi: 10.1007/s00404-009-1002-7. Epub 2009 Mar 7. PMID 19271230
- [Background] Bujold E, Roberge S, Lacasse Y, Bureau M, Audibert F, Marcoux S, Forest JC, Giguere Y. Prevention of preeclampsia and intrauterine growth restriction with aspirin started in early pregnancy: a meta-analysis. Obstet Gynecol. 2010 Aug;116(2 Pt 1):402-414. doi: 10.1097/AOG.0b013e3181e9322a. PMID 20664402
- [Background] Sealed Envelope Ltd. Power calculator for binary outcome equivalence trial. [Online]. 2012. Available from: https://www.sealedenvelope.com/power/binary-equivalence/.
- See also: Published PIPSICKLE TRIAL protocol — https://bmjopen.bmj.com/content/bmjopen/11/8/e047949.full.pdf

DOCUMENTS (2):
  • Study Protocol (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT05253781/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT05253781/SAP_001.pdf